CLINICAL TRIAL: NCT06703268
Title: A Multicenter, Randomized, Open-label, Controlled Study on Evaluating the Efficacy and Safety of Switching From Daily DPP-4 Inhibitors to HSK7653 Tablets in Patients With Type 2 Diabetes Mellitus in China
Brief Title: A Study on Switching From Daily DPP-4 Inhibitor to HSK7653 in Type 2 Diabetes Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK7653-203
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes
Keywords: HSK7653; DPP-4i
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK7653 (Experimental): HSK7653 10mg Q2W
  Interventions: Drug: HSK7653 10 mg
- Daily DPP-4 inhibitor (Active Comparator): Daily DPP-4 inhibitor
  Interventions: Drug: Daily DPP-4 inhibitor

INTERVENTIONS:
Drug: HSK7653 10 mg — HSK7653 10 mg Q2W
  Arms: HSK7653
Drug: Daily DPP-4 inhibitor — Daily DPP-4 inhibitor
  Arms: Daily DPP-4 inhibitor

SUMMARY:
To assess the effectiveness of HSK7653 tablets following the substitution of daily DPP-4 inhibitor (DPP-4i) over a 24-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and Age ≤75 years
* T2DM patients,
* During the 12 weeks before screening, on the basis of diet control and exercise therapy, patients only regularly received daily DPP-4 inhibitors (such as sitagliptin, vildagliptin, saxagliptin, linagliptin, alogliptin and retagliptin , etc.) or combined with metformin (with a metformin dose of ≥ 1500 mg/day, or the maximum tolerated dose < 1500 mg/day but ≥ 1000 mg/day);
* HbA1c ≥6.5% and HbA1c <8.0%
* FPG <10.0 mmol/L
* BMI ≥19 and BMI ≤ 35 kg/m2 (Body Mass Index)

Exclusion Criteria:

* Non-type 2 diabetes: Type 1 diabetes, gestational diabetes or other special types of diabetes.
* The presence of any of the following medical histories or conditions at the time of screening:
* History of diabetic ketoacidosis or hyperglycemic hyperosmolar state within the recent 6 months;
* History of ≥2 episodes of severe hypoglycemia within the last 6 months;
* History of malignant tumors within the recent 5 years (except for cured basal cell carcinoma of the skin and cervical carcinoma in situ), or currently being evaluated for potential malignant tumors.
* Presence of severe mental disorders or language barriers, unwilling or unable to fully understand and cooperate.
* History of drug abuse within the past 5 years
* Previous history or clinical evidence of acute or chronic pancreatitis.
* Using other drugs that may affect blood glucose metabolism within 12 weeks prior to screening, including systemic glucocorticoids (except for inhaled or topical ones), growth hormones, etc.
* Any laboratory test index meeting the following criteria:
* Hemoglobin < 110 g/L (for males) or < 100 g/L (for females).
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 3 times the upper limit of the normal value.
* Total bilirubin (TBIL) > 2 times the upper limit of the normal value.
* Fasting triglyceride (TG) > 5.7 mmol/L.
* Estimated glomerular filtration rate (eGFR) calculated using the CKD-EPI formula < 45 mL/min/1.73m².
* Known to be allergic to the investigational products or related excipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Time in range | 24 weeks
  The change in time in range (TIR) of continuous glucose monitoring (CGM) relative to the baseline after 24 weeks of treatment.

SECONDARY OUTCOMES:
HbA1c | 24 weeks
  Change from baseline in HbA1c after 24 weeks
Fasting glucose | 24 weeks
  Change from baseline in fasting glucose after 24 weeks
Mean glucose | 24 weeks
  Change from baseline in mean glucose after 24 weeks
Treatment-emergent adverse events. | 24 weeks
  The incidence of treatment-emergent adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Hsien-I Memorial Hospital, Tianjin Medical University, Tianjin, China

IPD SHARING:
Plan to Share IPD: No